CLINICAL TRIAL: NCT04991506
Title: An Open-label, Multicenter, Dose-escalation and Cohort Expansion Phase 1 Clinical Study of ES102 in Combination With JS001 in Patients With Advanced Solid Tumors
Brief Title: A Study of ES102 (OX40 Agonist) in Combination With JS001 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Elpiscience Biopharma, Ltd. (Industry)
Collaborators: Shanghai Junshi Bioscience Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ES102-1002
Record Dates: First submitted 2021-07-19; First posted 2021-08-05 (Actual); Last update posted 2025-06-23 (Actual); Status verified 2025-06

CONDITIONS: Solid Tumor; Neoplasms; Malignant Tumor
Keywords: ES102; JS001; OX40; PD-1; Solid Tumors; Phase 1; INBRX-106
MeSH Terms: conditions — Neoplasms | interventions — toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Part 1 ES102 Escalation in combination with JS001 (Experimental): ES102 will be escalated, in combination with JS001, in patients with advanced solid tumors.
  Interventions: Drug: ES102; Drug: JS001
- Part 2 ES102 Expansion in combination with JS001 (Experimental): Subjects will be treated with ES102 at the RP2D in combination with JS001.
  Interventions: Drug: ES102; Drug: JS001

INTERVENTIONS:
Drug: ES102 — The active ingredient of ES102 is a recombinant, humanized, hexavalent IgG antibody that targets the human OX40 receptor (TNFRSF4)
Drug: JS001 — JS001 is administered via intravenous injection once every 21 days, every 21 days as a treatment cycle.
  Other Names: Toripalimab

SUMMARY:
The purpose of this study is to evaluate the safety, tolerance, Dose-Limiting Toxicity (DLT), Maximum tolerated dose (MTD) and/or Recommended Phase 2 Dose (RP2D) of ES102 (OX40 agonist) in combination with JS001 (anti-PD-1 checkpoint inhibitor) in patients with advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* 1.Males or females aged ≥18 years.
* 2.Ability to understand and the willingness to sign a written informed consent form.
* 3.Subjects with pathological or cytological diagnosed advanced solid tumor, whose disease has progressed despite standard therapies, or for whom no further standard therapy exists, or who is unsuitable for available standard therapies and at least has progressed after receiving first line therapy.
* 4.PD-L1 by IHC: Parts 1 and Part 2 D2-D3: IHC result mandatory but any score allowed. Part 2 D1: Tumor Proportion Score (TPS) ≥ 1%.
* 5.At least one measurable lesion is required (RECIST v1.1)
* 6.Adequate hematologic, coagulation, hepatic and renal function as defined per protocol.
* 7.Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 or 1.
* 8.Estimated life expectancy, in the judgment of the investigator, of at least 12 weeks.
* 9.Male and female subjects of childbearing potential and their spouses must be willing to use feasible contraceptive methods considered effective by the investigator, from the time of signing informed consent and for the duration of study participation through 3 months, following the last dose of study drug. Postmenopausal women are considered to have no fertility potential only if menostasis lasts for at least 12 months.

Exclusion Criteria:

* 1.Prior exposure to OX40 agonists.
* 2.Receipt of any anticancer investigational product or any approved anticancer drug(s) or biological product(s) within 4 weeks prior to the first dose of study drug with certain exceptions.
* 3.Receipt of non-CNS adjuvant radiation therapy within 1 week prior to the first dose, receipt of radiation therapy within 2 weeks or with radiation pneumonia, have not recovered from radiation-related toxicity or still require hormonal treatment for radiation-related toxicity.
* 4.Known allergies to CHO-produced antibodies, which in the opinion of the Investigator suggests an increased potential for an adverse hypersensitivity to ES102.
* 5.Subjects with allergic reactions to the active ingredients of JS001 or any of the excipients.
* 6.Treatment with systemic immunosuppressive medications within 4 weeks prior to the first dose of study drug. Certain exceptions as defined in protocol apply.
* 7.Receipt of live viral vaccine treatment within 4 weeks prior to the first dose of the study drug.
* 8.Prior organ allograft transplantations or allogeneic peripheral blood stem cell (PBSC) or bone marrow (BM) transplantation.
* 9.Subjects with primary or metastatic brain or meningeal tumors.
* 10.Grade ≥ 3 immune-related adverse events (irAEs) or irAE that lead to discontinuation of prior immunotherapy. Some exceptions as defined per protocol apply.
* 11.Subject has not recovered from all AEs of previous anticancer therapies to baseline or ≤ Grade 1 per CTCAE v5.0 before the first dose of study drug. Certain exceptions as defined in protocol apply.
* 12.Hematologic malignancies.
* 13.Receipt of treatment with G-CSF, GM-CSF, Thrombopoietic drugs or EPO within 14 days prior to the first dose of the study drug.
* 14.Patients with other malignancies within 2 years before screening shall be excluded in Part B. Some exceptions as defined per protocol apply.
* 15.Active autoimmune disease or documented history of autoimmune disease that required systemic steroids or other immunosuppressive medications. Certain exceptions as defined in protocol apply.
* 16.Active interstitial lung disease (ILD) or pneumonitis or a history of ILD or pneumonitis requiring treatment with steroids or other immunosuppressive medications.
* 17.Clinically significant cardiac condition, including myocardial infarction, uncontrolled angina, cerebrovascular accident, or other acute uncontrolled heart disease < 6 months; left ventricular ejection fraction (LVEF) < 50%; New York Heart Association (NYHA) Class III or IV congestive heart failure; or uncontrolled hypertension.
* 18.History of pulmonary embolism within 12 weeks prior to the first dose of study drug administration.
* 19.Major surgery within 4 weeks prior to enrollment on this trial.
* 20.History of hepatitis B, hepatitis C, or human immunodeficiency virus (HIV) infection for Part 1. Exceptions as defined in protocol for Part 2 will apply.
* 21.Receiving the systemic anti-infectious drug treatments within 4 weeks prior to the first dose of study drug.
* 22.Pregnant or nursing females.
* 23.Any known, documented, or suspected history of substance abuse that would preclude subject from participation, certain exceptions as defined in protocol apply.
* 24.The subject is inappropriate to participate in this study for other reasons in the judgment of the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2024-05-17 (Actual); Study Completion 2024-05-17 (Actual)

PRIMARY OUTCOMES:
MTD | 2-4 years
  Maximum Tolerated Dose (MTD) of ES102 in combination with JS001
Frequency and severity of adverse events of ES102 in combination with JS001 | 2-4 years
  The safety profile of ES102 in combination with JS001 will be assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 5.0.
RP2D | 2-4 years
  Recommended Phase 2 Dose (RP2D) of ES102 in combination with JS001

SECONDARY OUTCOMES:
Area under the serum concentration time curve (AUC) of ES102 in combination with JS001 | 2-4 years
  Area under the serum concentration time curve (AUC) of ES102 in combination with JS001 will be determined.
Maximum observed serum concentration of ES102 in combination with JS001 | 2-4 years
  Maximum observed serum concentration of ES102 in combination with JS001 will be determined.
Trough observed serum concentration (Ctrough) of ES102 in combination with JS001 | 2-4 years
  Trough observed serum concentration (Ctrough) of ES102 in combination with JS001 will be determined.
Time to Cmax (Tmax) of ES102 in combination with JS001 | 2-4 years
  Time to Cmax (Tmax) of ES102 in combination with JS001 will be determined.
Immunogenicity of ES102 in combination with JS001 | 2-4 years
  Frequency of anti-drug antibodies (ADA) against ES102 in combination with JS001 will be determined.
Anti-tumor activity of ES102 in combination with JS001 | 2-4 years
  Tumor response will be determined by the revised Response Evaluation Criteria in Solid Tumors version 1.1 (RECISTv1.1).

CONTACTS AND LOCATIONS:
Locations (1):
- Jilin Cancer Hospital, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No